CLINICAL TRIAL: NCT05990075
Title: An eHealth Intervention to Increase Depression Treatment Initiation and Adherence Among Veterans Referred for Mental Health Services (CDA 18-189)
Brief Title: An eHealth Intervention to Increase Depression Treatment Initiation and Adherence Among Veterans Referred for Mental Health Services
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 21-002; IK2HX002899-01A2 (NIH)
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: depression; treatment initiation; treatment adherence; treatment utilization
MeSH Terms: conditions — Depression; Treatment Adherence and Compliance | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: The study employs a single group design given its focus on feasibility and acceptability.
Masking Description: The primary goal of the study is feasibility and acceptability of methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-monitoring (Experimental): This research study will evaluate a self-monitoring intervention to increase awareness, provide support, and promote motivation to initiate treatment after referral to mental health. The proposed intervention is a user-driven program delivered online and by mobile text. This will be initially piloted for acceptability among Veterans referred to mental health service for depression treatment.
  Interventions: Behavioral: self-monitoring

INTERVENTIONS:
Behavioral: self-monitoring — This research study will evaluate a self-monitoring intervention to increase awareness, provide support, and promote motivation to initiate treatment after referral to mental health. The proposed intervention is a user-driven program delivered online and by mobile text. This will be initially piloted for acceptability among Veterans referred to mental health service for depression treatment.

SUMMARY:
Depression is the most prevalent mental health condition among VHA patients and is strongly associated with poor functioning, negative health outcomes, and suicide. Despite effective and available treatments, engagement in care is poor. This study will analyze VHA electronic medical record data, to identify patient characteristics associated with poor treatment engagement. The study will then develop and formatively evaluate an eHealth intervention to improve and sustain engagement in mental health care through self-monitoring. This is an important step in engaging Veterans who, in part, based on their military training, may have difficulty identifying or accepting depressed affect and the benefits of treatment. The information obtained will inform clinical strategies and operations policy to improve quality, coordination, and efficiency of mental health services.

DETAILED DESCRIPTION:
My goal is to optimize treatment outcomes for Veterans with depression. To experience positive outcomes, Veterans must begin care promptly when needed and remain engaged in care. Depression imposes a great burden of illness and disability for the OEF/OIF Veteran population. As few as 30% of Veterans initiate treatment after referrals for mental health services and adherence after initiation is low. Untreated depression is strongly linked to suicide mortality, drug abuse, and persistent impairment leading to poor health outcomes. The VHA has focused on increasing access to evidence-based treatments (EBTs) as the gold standard for treating depression, however the guidelines do not address Veterans who are lost to care. This is a missed opportunity to engage Veterans who fail to initiate traditional treatment or drop out early, often due to discomfort and lack of awareness of certain depression symptoms or need for care, which translates to reduced self-efficacy to engage. Furthermore, measurement-based care-the utilization of systematic symptom assessments over time to drive changes in treatment-is recommended for care in VHA. Patients at risk for dropping out of care may find systematic assessments acceptable and effective for supporting engagement in EBTs if their symptoms persist.

This study addresses treatment initiation and adherence among depressed Veterans who are referred to mental health care. Specifically, the investigators will test an innovative self-monitoring program for Veterans with depression which has the potential to facilitate both treatment uptake and sustained engagement. The proposed research will test a patient centered, self-monitoring eHealth intervention focused on systematic measurement and feedback for Veterans with depression, as well as supportive messages providing VA related information and coping strategies that Veterans elect.

The intervention will be initiated when patients are referred for care. This program will continue to help Veterans monitor during treatment if they so desire, as self-monitoring has been found to increase the likelihood of treatment response. The objectives of this study are to formatively evaluate this process and provide preliminary support to then evaluate the efficacy/effectiveness of this intervention in a future study.

This project is aligned with the VHA HSR&D priorities in mental health and improving access to care and high-priority research topics for mental and behavioral health. Findings from this study have the potential to lead to transdiagnostic research, especially for PTSD, TBI, and suicide.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* Recent referral to VA general mental health clinics providing psychotherapy for depression
* No gender or minorities will be excluded from this study
* 18-64 will be included

Exclusion Criteria:

* Current/Past Bipolar disorder and Current Psychotic disorder: to avoid potential exacerbation from treatment for depression
* Alcohol Use disorder or Substance Use disorder: Depression treatments cannot reverse the adverse effects of substances on mood, and therefore impact on adherence and treatment characteristics may be confounded
* Other current severe or unstable, psychiatric and medical disorders that necessitates clinical management that can confound results (e.g., cancer [in chemotherapy], suicidality, recent hospitalization [medical/surgical] for which recovery overlaps with study onset and duration, open skull/brain injury, moderate to severe TBI)
* Moderate to severe cognitive impairment (SLUMS 20 and/or diagnosis in medical record)
* Potentially temporary states/situations that may significantly impair mood/capability to engage in treatment: unstable environment that is not in one's control (e.g., homeless, temporary group home, extensive care taking duties)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Panaite, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referrals to specialty mental health clinics for depressive disorders and depressive symptoms between September 2023-September 2024. Prior to enrollment, participant clinical charts were screened.
Pre-assignment Details: Of those who met inclusion criteria, 47 patients agreed to participation and enrolled in the study.
Period: Overall Study
Arm/Group | Self-monitoring
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Self-monitoring
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 14
  White | 22
  More than one race | 0
  Unknown or Not Reported | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 4
Marital status [Count of Participants; unit: Participants]
  Divorced | 11
  Married | 21
  Never Married | 11
  Separated | 3
  Unknown | 1
Service Connected (%) [Count of Participants; unit: Participants]
  0% | 4
  10-50% | 5
  60-90% | 17
  100% | 21
Service Connected for Mental Health [Count of Participants; unit: Participants]
  Yes | 33
  No | 14
Barriers to Accessing Care Evaluation (BACE) [Mean (Standard Deviation); unit: Units on a scale] — BACE is a comprehensive measure that identifies stigma, access, and practical barriers individuals face when seeking mental health. Items are scored on a 0 (Not at all) to 3 (A lot) scale.
  Units on a scale
    Stigma related barriers | 0.64 (0.50)
    Access and practical barriers | 1.04 (0.50)
Affective Control Scale (ACS) [Mean (Standard Deviation); unit: Units on a scale] — ACS measures fear of losing control over one's negative and positive emotions or of one's behavioral reactions to these emotions. Items are scores on a 1 (Very Strongly Disagree) to 7 (Very Strongly Agree) scale.
  Units on a scale
    Fear of anger | 4.20 (1.11)
    Fear of positive emotions | 3.47 (0.91)
    Fear of depression | 4.19 (0.97)
    Fear of anxiety | 4.39 (1.05)
Patient Health Questionnaire 8 (PHQ8) [Mean (Standard Deviation); unit: Units on a scale] — PHQ8 assesses depression related symptoms on a 0 = Not at all 1 = Several days 2 = More than half the days 3 = Nearly every day scale. Scores range from 0 to 24 with higher scores indicating higher depression symptoms.
  Units on a scale | 15.34 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Intervention Enrollment as Assessed by Completion of Baseline Survey.
Description: Intervention enrollment was measured by completion of baseline survey which entailed patients' explicit agreement to participate in the intervention.
Time Frame: Up to 30 weeks.
Population: The denominator for this analysis were participants who were pre-screened, met study criteria, and were invited to participate in the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-monitoring
Number analyzed (Participants) | 270
Participants | 47

2. Primary Outcome: Percent Patients With Completed Tasks as Measured by Mental Health Link.
Description: Mental Health Link asks patients to report on 24 hour positive and negative events, emotions, and depression symptoms.
Time Frame: Immediately after intervention completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-monitoring
Number analyzed (Participants) | 47
Participants
  Engagement with intervention | 47
  > 50% engagement rate | 25

3. Other Pre Specified Outcome: Efficacy of Intervention as Assessed by Rate of Depression Treatment Initiation and Adherence
Description: The investigators will evaluate % mental health treatment initiation relative to the general population in the same clinics. This measure is experimental given that efficacy is not yet the focus of this work given its preliminary stage. Treatment initiation is defined as initial mental health appointment being completed. Treatment adherence is defined as continuing treatment past initiation.
Time Frame: Immediately after intervention, up to 30 weeks.
Population: Denominator for treatment adherence is number of patients who initiated treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-monitoring
Number analyzed (Participants) | 47
Participants
  Treatment initiation | 32
  Treatment adherence (1+ sessions): number analyzed (Participants) | 32
  Treatment adherence (1+ sessions) | 28
  Treatment adherence (4+ sessions): number analyzed (Participants) | 32
  Treatment adherence (4+ sessions) | 18

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 12 months
Arm/Group | Self-monitoring
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

LIMITATIONS AND CAVEATS:
This is a pilot study of an experimental technology based tool designed to help patients stay engaged after referral to mental health services. Sample size limits power for more complex analyses. Furthermore patients were allowed to engage with this tool as needed, and therefore data collected over time is highly variable, contributing to limitations for data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT05990075/Prot_001.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT05990075/SAP_002.pdf
  • Informed Consent Form (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT05990075/ICF_000.pdf